CLINICAL TRIAL: NCT06925984
Title: The Oligopro-Breast Study: Stereotactic Radiotherapy for Oligoprogressive ER+/HER- Metastatic Breast Cancer, a Prospective Phase 2 Study
Brief Title: Stereotactic Radiotherapy for Oligoprogressive ER+/HER- Metastatic Breast Cancer, a Prospective Phase 2 Study (Oligopro-Breast)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE4005
Record Dates: First submitted 2025-03-26; First posted 2025-04-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: OligoProgressive Metastatic Disease
Keywords: Oligoprogression; metastatic breast cancer; CDK4/6 inhibitors; SBRT; SABR; radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT on the oligoprogressive metastases. Continuation of same systemic therapy. (Experimental)
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT of all oligoprogressive metastases (or other local therapy if SBRT not advisable), followed by continuation of the same systemic therapy.

SUMMARY:
The Oligopro-Breast trial is a Phase II study targeting women with ER+/HER2- metastatic breast cancer who have been on endocrine therapy and/or CDK4/6 inhibitors for at least 6 months, and show progressive disease at 1-3 extracranial metastases, which are treatable locally. The trial aims to investigate if treating these resistant metastases with SBRT (or other local treatments if SBRT is not possible) can extend the use of the current systemic therapy.

Patients will continue their existing systemic treatment while receiving SBRT on all progressive lesions. If new oligoprogression occurs, SBRT will be performed again. A new systemic treatment line will start if there is polyprogression (more than 3 lesions at once), progression of more than 6 lesions over 12 months, intracranial progression, or lesions that cannot be treated locally.

The scientific question is whether local treatment of resistant metastases can prolong the effectiveness of ongoing systemic therapy, which is particularly beneficial if the treatment is well-tolerated. The primary objective is to measure the proportion of patients surviving without changing their systemic treatment line at 6 months after SBRT.

This trial is significant for patients as it explores a method to potentially extend the duration of effective and well-tolerated treatments, offering hope for better management of metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2.
* Histologically confirmed ER+/HER2- MBC.
* History of polymetastatic disease. Patients with genuine oligometastatic disease and 1-3 oligoprogressive lesions are only allowed if ablative therapy of all metastases is deemed impossible.
* Under 1st to 2nd systemic treatment line with hormonotherapy and/or CDK4/6 inhibitors for at least 6 months before progression.
* Progressive disease at 1-3 extracranial sites.
* Ability to treat all progressive lesions locally according to the treating radiation oncologist.

Exclusion Criteria:

* Second malignancy if it is not in complete remission.
* Previous local treatment for oligoprogression under the current systemic treatment line
* Current progression in a lesion that has been treated with SBRT before and is not amendable for surgery or radiofrequency ablation (RFA).
* Progressive or newly diagnosed brain metastases. Known brain metastases that have been nonprogressive for at least 6 months, are not an exclusion criterion.
* Inability to continue the same ST line after local therapy (for example because of toxicity or patient refusal).
* Pregnancy.
* Inability to sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
NExt Systemic Treatment-Free Survival (NEST-FS) | At 6 months

SECONDARY OUTCOMES:
Time to next line of systemic therapy (NEST) | 3 years
Progression-free survival (PFS) | 3 years
Modified Progression-free survival (mPFS) | 3 years
  Defined as the survival in the absence of any of the following : (1) polyprogression (progressive disease of more than 3 lesions at the same time), (2) progression of more than 6 lesions over a 12-month rolling period, (3) intracranial progression, (4) progressing lesion that cannot be treated locally, or (5) death.
Chemotherapy-free survival | 3 years
Progression-free survival after start of the subsequent line of systemic treatment (PFS2) | 3 year
Patterns of metastatic progression | 3 years
  We defined four patterns of progression: stable disease, progression on untreated pre-existing lesions, progression on treated lesions, or development of new lesions. In case of progression, it will also be determined whether it is oligoprogression (progression of 3 lesions or less) or polyprogression (progression of more than 3 lesions).
Overall survival (OS) | 3 years
Acute and late physician-scored toxicity of the local intervention | 3 years
  Acute and late physician-scored toxicity of the local intervention (CTCAE 5.0, Early: within 90 days; late: 90 or more days after SBRT);
Quality of life (QoL) | 3 years
  Evolution of QoL measured with the EORTC QLQ-C30

OTHER OUTCOMES:
Correlation between (1) ctDNA burden at baseline and (2) ctDNA burden 10-12 weeks after SBRT versus the modified progression-free-survival (mPFS). NEST-FS in function of ESR1 status. | 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - Jules Bordet Institute, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - AZ Sint-Maarten, Mechelen
  - CHU UCL Namur - Site Saint Elisabeth, Namur

IPD SHARING:
Plan to Share IPD: No